CLINICAL TRIAL: NCT06975176
Title: Combating HIV Stigma in Healthcare Settings: A Standardized Patient Approach
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIV Stigma
Record Dates: First submitted 2025-03-18; First posted 2025-05-16 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Hiv
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stigma Reduction Intervention (Experimental): A Stigma Reduction Intervention curriculum developed using data generated from Stage 1 of the study.
  For stage 2/intervention stage, participants who are providers and randomized to the "Stigma Reduction Intervention" arm through clinic-level randomization
  Interventions: Behavioral: Stigma reduction intervention
- Control (No Intervention): For stage 2/intervention stage, participants who are providers and randomized to the "Control" arm through clinic-level randomization

INTERVENTIONS:
Behavioral: Stigma reduction intervention — Care providers will complete the Stigma Reduction Intervention curriculum. The intervention is a multi-day stigma reduction training program for providers.
  Content design is greatly informed by materials developed in our pilot R34 study, and which may be modified prior to the intervention if the team gains new insights from the baseline round of unannounced visits and each of the two CABs. Briefly, the intervention consists of both didactic and experiential learning components. Didactic sessions include instruction on syphilis epidemiology, clinical management, and public health significance. Experiential sessions include discussion sessions that are facilitated by pre-recorded videos, followed by role play with trained SPs.
  Arms: Stigma Reduction Intervention

SUMMARY:
The goal of this study is to develop and evaluate the effectiveness of a training program to reduce intersectional stigma faced by sexual minorities and people living with HIV (PLWH) in healthcare settings. The study participants are medical providers (i.e. physicians) specializing in sexual health medicine in China.

DETAILED DESCRIPTION:
Consistent data highlight the central role of stigma in limiting uptake of HIV related testing, treatment, and care. This is particularly true for gay, bisexual, and other MSM who have the lowest rates of engagement with the healthcare system despite bearing the highest HIV incidence burden. Particularly for MSM seeking HIV testing services, enacted stigma-overt acts of discrimination and hostility directed at a person because of their perceived stigmatized status -both on account of their same-sex behaviors (i.e. sexuality stigma or homophobia) and the perception of their elevated HIV risk (HIV stigma) is all too common. Trained standardized patients (SP) will present a standardized case to providers.

SPs will present clinically standardized case scenarios, but the HIV status and sexual orientation of each case will be randomly varied. Stigma will be evaluated by comparing the quality of care that SPs experience during provider visits. Results of the baseline visit will inform the development of a stigma reduction training program for provider participants employed at clinics randomized to the treatment arm. The overall structure consists of didactic content as well as experiential learning using simulation-and-feedback sessions with trained SPs.

ELIGIBILITY:
Inclusion Criteria:

Eligible facilities are those with

* formal government accreditation as a medical center (a basic tenet of all public hospitals in China); and
* possession of an accredited on-site laboratory with capacity to provide enzyme- linked immunosorbent assay testing for HIV, treponemal (e.g. Treponema pallidum particle agglutination) and non-treponemal tests (e.g. rapid plasma regain) for syphilis. Within eligible and consenting facilities, eligible providers are those who are licensed at the time of the study to practice STD care in China.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Impact of the intervention on healthcare stigma directed at men who have sex with men (i.e. homophobia) in which stigma is measured as differences in whether or not syphilis testing was offered to MSM vs straight patients. | 3 months
  The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. This outcome compares pre-post changes in MSM stigma across study arms (i.e. differences in care quality between men who have sex with men [MSM] vs. straight men). This particular outcome measures care quality in terms of whether or not doctors offered a syphilis test.
Impact of the intervention on healthcare stigma directed at people living with HIV (i.e. HIV stigma), in which stigma is measured as differences in whether or not syphilis testing was offered to patients living with HIV vs those not living with HIV. | 3 months
  The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. This outcome compares pre-post changes in HIV stigma across study arms (i.e. differences in care quality between people living with HIV [PLWH] vs. those who are not living with HIV). This particular outcome measures care quality in terms of whether or not doctors offered a syphilis test.
Impact of the intervention on healthcare stigma directed at people living with HIV who are also MSM (i.e. intersectional stigma), measured as differences in whether syphilis testing was offered to MSM with HIV vs. straight men without HIV. | 3 months
  The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. This outcome compares pre-post changes in intersectional stigma across study arms (i.e. differences in care quality between MSM living with HIV vs. straight men not living with HIV). This outcome measures care quality related to whether or not doctors offered a syphilis test. This particular outcome measures care quality in terms of whether or not doctors offered a syphilis test.
Impact of the intervention on healthcare stigma directed at men who have sex with men (i.e. homophobia), in which stigma is measured as differences in the level of diagnostic effort expended by doctors for MSM patients vs straight patients. | 3 months
  The outcome represents the amount by which stigma was reduced in each arm between baseline and follow-up. Stigma itself was measured as the difference in healthcare quality between a stigmatized group vs. a dominant group. Because healthcare is multidimensional, we examined it across three domains: syphilis testing, diagnostic effort, and patient-centeredness of care. Positive values mean stigma indicate a decrease in stigma between the two time points. Negative values mean an increase in stigma between the two time points. This outcome compares pre-post changes in MSM stigma across study arms (i.e. differences in care quality between men who have sex with men [MSM] vs. straight men). This particular outcome measures care quality in terms of the level of diagnostic effort expended. Our measure of diagnostic effort is a composite indicator constructed from 18 items relating to various aspects of diagnostic care such as history taking and physical examinations.
Impact of the intervention on healthcare stigma directed at people living with HIV (HIV stigma), in which stigma is measured as differences in diagnostic effort expended by doctors for patients living with HIV vs. patients not living with HIV. | 3 months
  The outcome reflects the amount by which stigma was reduced in each arm between baseline and follow-up. Stigma was measured as the difference in healthcare quality between stigmatized and dominant groups. Because healthcare is multidimensional, we examined three domains: syphilis testing, diagnostic effort, and patient-centeredness. Positive values indicate decreased stigma; negative values indicate increased stigma. This outcome compares pre-post changes in HIV stigma across study arms (i.e. differences in care quality between people living with HIV [PLWH] and those not living with HIV). It measures care quality by the level of diagnostic effort. Diagnostic effort is a composite indicator based on 18 items on history taking, physical exams, and other aspects of care. The scale was developed by the study team using Chinese clinical guidelines and input from local physicians experienced in person-centered sexual health care. Items use 4-point Likert scales summed into a provider score.
Impact of the intervention on healthcare stigma directed at people living with HIV and who are MSM (i.e. intersectional stigma), in which stigma is measured as differences in diagnostic effort by doctors for MSM with HIV vs. straight men without HIV. | 3 months
  The outcome reflects how much stigma was reduced in each arm between baseline and follow-up. Stigma was measured as the difference in healthcare quality between stigmatized and dominant groups. As healthcare is multidimensional, we examined three domains: syphilis testing, diagnostic effort, and patient-centeredness. Positive values indicate a decrease in stigma between time points; negative values indicate an increase. This outcome compares pre-post changes in intersectional stigma across study arms (i.e. differences in care quality between MSM with HIV and HIV-negative straight men). It measures care quality by level of diagnostic effort. Diagnostic effort is a composite indicator based on 18 items covering history taking, physical exams, and other aspects of care. The scale was developed by the study team using Chinese clinical guidelines and input from local physicians experienced in person-centered sexual health care. Items use 4-point Likert scales, summed into a provider score.
Impact of the intervention on healthcare stigma directed at men who have sex with men (homophobia), in which stigma is measured as differences in the patient-centeredness of care provided to MSM vs. straight patients. | 3 months
  The outcome reflects how much stigma was reduced in each arm between baseline and follow-up. Stigma was measured as the difference in healthcare quality between stigmatized and dominant groups. As healthcare is multidimensional, we examined three domains: syphilis testing, diagnostic effort, and patient-centeredness. Positive values indicate a decrease in stigma between time points; negative values indicate an increase. This outcome compares pre-post changes in MSM stigma across study arms (i.e., differences in care quality between MSM and straight men). It specifically measures care quality in terms of patient-centeredness. Our measure of patient-centeredness is a composite indicator based on 19 items like doctors' word choice and use of nonverbal communication. The scale was developed by the study team using Chinese clinical guidelines and input from local physicians experienced in person-centered sexual health care. Items use 4-point Likert scales, summed into a provider score.
Impact of the intervention on healthcare stigma directed at people living with HIV (HIV stigma), in which stigma is measured as differences in the patient-centeredness of care provided to patients living with HIV vs. those not living with HIV. | 3 months
  The outcome reflects how much stigma was reduced in each arm between baseline and follow-up. Stigma was measured as the difference in healthcare quality between a stigmatized group and a dominant group. As healthcare is multidimensional, we examined three domains: syphilis testing, diagnostic effort, and patient-centeredness. Positive values indicate a decrease in stigma; negative values indicate an increase. This outcome compares pre-post changes in HIV stigma across study arms (i.e., differences in care quality between people living with HIV [PLWH] and those not living with HIV). It specifically measures care quality based on patient-centeredness. Our measure is a composite indicator from 19 relevant items such as doctors' word choice or nonverbal communication. The scale was developed by the study team using Chinese clinical guidelines and input from local physicians experienced in person-centered sexual health care. Items use 4-point Likert scales, summed into a provider score.
Impact of the intervention on healthcare stigma directed at people living with HIV and who are MSM (i.e. intersectional stigma), in which stigma is measured as differences in patient-centeredness of care for MSM with HIV vs. straight men without HIV. | 3 months
  The outcome reflects how much stigma was reduced in each arm between baseline and follow-up. Stigma was measured as the difference in healthcare quality between stigmatized and dominant groups. As healthcare is multidimensional, we examined three domains: syphilis testing, diagnostic effort, and patient-centeredness. Positive values indicate a decrease in stigma; negative values indicate an increase. This outcome compares pre-post changes in intersectional stigma across study arms (i.e. differences in care quality between MSM with HIV and straight men without HIV). It specifically measures care quality based on patient-centeredness. Our measure is a composite indicator constructed from 19 items such as doctors' word choice or use of nonverbal communication. The scale was developed by the study team using Chinese clinical guidelines and input from local physicians experienced in person-centered sexual health care. Items use 4-point Likert scales, summed into a provider score.

CONTACTS AND LOCATIONS:
Overall Officials: Kumi Smith, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States